CLINICAL TRIAL: NCT05851027
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Phase 3 Study Evaluating the Efficacy and Safety of Recombinant Human Thrombopoietin Mimetic Peptide-Fc Fusion Protein for Injection (QL0911) in Chemotherapy- Induced Thrombocytopenia
Brief Title: Evaluating the Efficacy and Safety of QL0911 in Chemotherapy- Induced Thrombocytopenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL0911-CIT-301(PartA）
Record Dates: First submitted 2023-04-23; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Chemotherapy-induced Thrombocytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QL0911 Group 1 (Experimental): Starting dose 1μg/kg；PLT 100~200×10^9/L
  Interventions: Drug: QL0911
- QL0911 Group 2 (Experimental): Starting dose 2μg/kg；PLT 100~200×10^9/L
  Interventions: Drug: QL0911
- QL0911 Group 3 (Experimental): Starting dose 2μg/kg；PLT <100×10^9/L
  Interventions: Drug: QL0911

INTERVENTIONS:
Drug: QL0911 — Qilu investigational product (QL0911 or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.

SUMMARY:
To evaluate the efficacy and safety of QL0911 in Chemotherapy- Induced Thrombocytopenia. Thrombocytopenia is a low number of platelets in the blood. Sometimes, thrombocytopenia is a side effect of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old when signing the informed consent form;
* Histopathological or cytological examination, confirmed as solid tumor or lymphoma (including NSCLC, breast cancer, bladder cancer, pancreatic cancer, etc.), the chemotherapy cycle is 21 days or 28 days, and one or more of the following chemotherapy drugs are needed: anti-metabolic drugs, including gemcitabine, etc.; Platinum, including carboplatin, nedaplatin, cisplatin, lobaplatin, etc. Anthracyclines, including adriamycin, daunorubicin, epirubicin, etc. Alkylating agent, including cyclophosphamide, ifosfamide, etc. Other cytotoxic chemotherapy drugs that can cause thrombocytopenia;
* In the last regular chemotherapy cycle, the subject had a decrease in platelet count below 75× 109/L;
* Platelet count ≤ 200× 109/L one day before chemotherapy;
* The estimated survival time at screening is ≥12 weeks, and the current chemotherapy regimen can be accepted for at least 2 cycles (at least 1 cycle in PartA);
* According to the score standard of physical fitness of the Eastern Cancer Cooperative Group (ECOG), it is 0-2;
* Fully understand and abide by the requirements of this study, and sign the informed consent form voluntarily.

Exclusion Criteria:

* Suffering from other hematopoietic diseases except lymphoma, including leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma and myelodysplastic syndrome;
* Thrombocytopenia caused by non-tumor chemotherapy drugs occurred within 6 months before screening, including but not limited to EDTA-dependent pseudothrombocytopenia, hypersplenism, infection and bleeding;
* Bone marrow invasion or bone marrow metastasis occurs;
* Being receiving radiotherapy or having received abdominal or pelvic radiotherapy within 3 months;
* There have been any arterial or venous thrombosis events within 6 months before screening;
* Screening patients with severe cardiovascular disease (NYHA cardiac function score III-IV) and arrhythmia that increases the risk of thrombosis, such as atrial fibrillation, after coronary stent implantation, angioplasty and coronary artery bypass grafting;
* Clinical manifestations of severe bleeding (such as gastrointestinal bleeding, etc.) within 2 weeks before screening;
* Received platelet transfusion within 2 days before randomization;
* Patients have been treated with thrombopoietin receptor agonists (such as romistine and itrapoppa) or human recombinant thrombopoietin (rhTPO) or rhIL-11 within 4 weeks before the first administration;
* Anticoagulant drugs such as heparin, warfarin and aspirin have been used within 7 days before the first administration;
* Received bone marrow transplantation or stem cell infusion within one year before screening;
* Patients with chronic hepatitis B or hepatitis C in active period, and patients with positive antibodies to human immunodeficiency virus;
* The absolute value of neutrophils in the screening period is less than 1.5× 109/L, and hemoglobin is less than 90g/L;
* The total bilirubin in the screening period is more than 3 times the upper limit of the normal range; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were higher than the upper limit of normal range by 3 times. For patients with liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≥ 5 times the upper limit of the normal range;
* Blood creatinine concentration ≥1.5ULN or EGFR ≤ 60 ml/min;
* patients with severe drug allergic reaction;
* Patients who have used any research drugs (excluding vitamins and minerals) within 3 months before the first administration;
* Patients who plan pregnancy, pregnancy or lactation;
* The researcher judges the patients who are not suitable for this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
The effective response rate of QL0911 on the 21st day (21-days chemotherapy cycle) after administration. | 21 days
The effective response rate of QL0911 on the 28th day (28-days chemotherapy cycle) after administration. | 28 days

SECONDARY OUTCOMES:
Changes of platelet count from baseline in each visit(21-days chemotherapy cycle) | 21 days
Changes of platelet count from baseline in each visit(28-days chemotherapy cycle) | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China